CLINICAL TRIAL: NCT00006000
Title: Phase I Study of SU5416 in Combination With CPT-11 and Cisplatin in Patients With Solid Tumors
Brief Title: SU5416, Irinotecan, and Cisplatin in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068008; OSU-00H0033; NCI-47
Record Dates: First submitted 2000-07-05; First posted 2004-03-05 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2002-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; Irinotecan; Semaxinib

INTERVENTIONS:
Drug: cisplatin
Drug: irinotecan hydrochloride
Drug: semaxanib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. SU5416 may stop the growth of solid tumors by stopping blood flow to the tumor. Combining SU5416 with chemotherapy may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of SU5416 plus irinotecan and cisplatin in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of SU5416 in combination with irinotecan and cisplatin in patients with advanced solid tumors. II. Determine the quantitative and qualitative toxicity of this treatment regimen in terms of organ specificity, time course, predictability, and reversibility in this patient population. III. Determine the therapeutic response of this treatment regimen in these patients. IV. Evaluate the clinical pharmacokinetics and the relationship of kinetics to toxicity and response in this patient population treated with this regimen.

OUTLINE: This is a dose escalation study of SU5416. Patients receive cisplatin IV over 90 minutes immediately followed by irinotecan IV over 90 minutes and SU5416 IV over 2 hours on day 1. Patients receive SU5416 alone on day 4. Patients receive combination chemotherapy weekly for 4 weeks and SU5416 twice weekly for 6 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of SU5416 until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced solid tumor for which no curative therapy exists No prior or concurrent primary brain tumor or brain metastasis

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-1 Life expectancy: At least 12 weeks Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 No inherited predisposition to hypercoagulation Hepatic: Bilirubin normal SGOT no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No uncompensated coronary artery disease on electrocardiogram or physical examination No myocardial infarction or severe unstable angina within the past 6 months No severe peripheral vascular disease related to diabetes mellitus No deep venous or arterial thrombosis within the past 3 months No inherited predisposition to thrombosis Pulmonary: No pulmonary embolism within the past 3 months Other: No other malignancies within the past 5 years except basal or squamous cell skin cancer or carcinoma in situ of the cervix No other significant medical illness No serious active infections Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy and recovered No concurrent biologic therapy Chemotherapy: At least 4 weeks since prior chemotherapy and recovered No other concurrent chemotherapy No prior cisplatin or irinotecan Endocrine therapy: At least 4 weeks since prior hormonal therapy and recovered No concurrent hormonal therapy Radiotherapy: At least 4 weeks since prior radiotherapy to less than 25% bone marrow and recovered No concurrent radiotherapy Surgery: At least 4 weeks since prior surgery and recovered No concurrent surgery Other: No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric H. Kraut, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio, United States